CLINICAL TRIAL: NCT02911766
Title: Comparing the Effect of 0,06 % -, 0,12 % and 0,2 % Chlorhexidine on Plaque, Bleeding and Side Effects in an Experimental Gingivitis Model. A Parallel, Double Masked, Randomized, Placebo-controlled Clinical Trial
Brief Title: Efficacy of Different Chlorhexidine Concentrations
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Hans Ragnar Preus, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2015/608453
Record Dates: First submitted 2016-09-09; First posted 2016-09-22 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Dental Plaque; Gingivitis
Keywords: Periodontal Index
MeSH Terms: conditions — Dental Plaque; Gingivitis | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Corsodyl, 0.2% mouthrinse (Active Comparator): The comparator solution was Corsodyl, 0.2% Chlorhexidine mouthrinse,
  Intervention Rinsing 60 sec with Comparator solution twice daily for 21 days
  Interventions: Drug: Chlorhexidine 0.2% Mouthrinse
- FluxProKlorhexidine 0.12% mouthrinse (Experimental): The experimental solution was FluxProChlorhexidine 0.12% mouthrinse
  Intervention Rinsing 60 sec with test solution twice daily for 21 days
  Interventions: Drug: Chlorhexidine 0.12% mouthrinse
- Corsodaily 0.06% mouthrinse (Experimental): The second experimental solution was Corsodaily, 0.06% chlorhexidine mouthrinse.
  Intervention Rinsing 60 sec with test solution twice daily for 21 days
  Interventions: Drug: Chlorhexidine 0.06% mouthrinse

INTERVENTIONS:
Drug: Chlorhexidine 0.2% Mouthrinse — Intervention; Rinsing 60 sec with Comparator solution twice daily for 21 days
  Other Names: Corsodyl 0.2% Chlorhexidine mouthwash
  Arms: Corsodyl, 0.2% mouthrinse
Drug: Chlorhexidine 0.12% mouthrinse — Intervention; Rinsing 60 sec with Comparator solution twice daily for 21 days
  Other Names: FluxProChlorhexidine 0.12%
  Arms: FluxProKlorhexidine 0.12% mouthrinse
Drug: Chlorhexidine 0.06% mouthrinse — Intervention; Rinsing 60 sec with Comparator solution twice daily for 21 days
  Other Names: Corsodaily 0.06% chlorhexidine mouthwash
  Arms: Corsodaily 0.06% mouthrinse

SUMMARY:
Chlorhexidine is the gold standard of dental plaque prevention, but which concentration is the most effective is not known. The aim of the present study was to compare the plaque and gingivitis inhibiting effect of commercial products containing 0.2%, 0.12% and 0.06% chlorhexidine in a modified experimental gingivitis model.

In three groups of healthy volunteers, experimental gingivitis was induced and monitored over 21days, simultaneously treated with the commercial solutions containing 0.2%, 0.12% and 0.06% chlorhexidine. The maxillary right quadrant of each individual received mouthwash only, whereas the maxillary left quadrant was subject to both rinsing and mechanical oral hygiene. Compliance and side effects were monitored at days 7, 14, and 21. Plaque and gingivitis scores were obtained at baseline and day 21.

The commercial mouthwash containing 0.2% chlorhexidine resulted in statistically significantly lower plaque scores than the 0.12 and 0.06% mouthwashes after 21 days use, whereas no statistically significant difference was found between the effect of the two latter mouthrinses.

A commercial available mouthwash containing 0.2% chlorhexidine proved statistically significant better effect in preventing dental plaque than 0.12% and 0.06% solutions.

DETAILED DESCRIPTION:
The present study was designed as a parallel, double masked, randomized, placebo-controlled clinical trial. The experimental gingivitis model, with the modifications by Preus and coworkers was used to induce gingival inflammation under supervised conditions throughout the study.

The study population comprised sixty dental, medical, and dental hygienist students who volunteered to participate in the project. A meeting was arranged for the volunteers prior to the start of the study, through which the participants received information about oral rinsing products in general and chlorhexidine containing products as well as information on the study ahead, in particular.

The study period was 21 days, not comprising any special academic, religious or ethnic events that could jeopardize the collective behavior of the study population. All information, administration and data collection was performed at the Department of Periodontology, Institute of Clinical Odontology, Faculty of Dentistry, University of Oslo, Norway.

The test solutions were the commercially available mouthwash products: 0.2 % chlorhexidine (no ethanol), 0.12% chlorhexidine with 910 ppm Sodium Fluoride (NaF) without ethanol and 0.06% chlorhexidine 250ppm Sodium Fluoride (NaF). The three commercially available chlorhexidine solutions were filled in identical, but differently labelled (A,B,C) plastic bottles for blinding purposes.

Randomization was carried out using a computer generated random allocation table, assigning the participants to the three study groups with 20 test subjects in each. They were all carefully instructed to rinse for 60 sec. twice a day as recommended by the manufacturers.

Setting the baseline dental plaque score to zero was done by giving all participants a professional tooth cleaning with rubber cup, pumice paste and dental floss at the start of the study. The participants were given their test solution and subsequently instructed to rinse as described above. All information was given verbally as well as in writing.

Individual plastic tooth guards had been produced to fit the teeth in the upper right quadrant. Together with this individual tooth guard, the students were given identical prophylaxis packs containing a medium texture tooth brush, inter-dental floss and dentifrice. The participants were instructed to substitute their daily oral hygiene remedies with the ones given to them, and attach the tooth guard to the tooth brush, with a provided rubber string, before and after use so that the use of this always was remembered when using the brush.

The participants were instructed to insert the tooth guard in the first quadrant every time they brushed their teeth and to perform a mechanical oral hygiene routine twice daily in the three other quadrants. They should then rinse 30 sec with tap water before and after removing the tooth guard to remove as much as possible of the remnants of the dentifrice. Following this procedure, the participants rinsed, as instructed, with the solution they randomly had been assigned, repeating the procedure for 21 days. Following the scoring at day 21, the participants received professional tooth cleaning after ending the study.

A team of five people were trained in the procedure of informing participants, receiving the test persons for evaluation, questionnaire and clinically monitoring them. The principal investigator and project managers managed all contact with the participants outside the scoring room. In between appointments the project team kept in touch with the test persons by text messaging and e-mail. The success of this service was evident by zero no-shows at the clinic, as was the case also in the previous studies with this design.

At the interviews at day 7, 14, 21 the project managers received reports from each participant about compliance (adherence to protocol) and verbal complaints and descriptions of subjective side-effects. A special questionnaire had been prepared for these interviews. Reports of ill- and side effects were carefully registered and categorized for later statistical examination.

At day 21, the above mentioned interview was followed by an examination of clinical results. Before entering the scoring room the project managers advised the participants to refrain from any conversation with the scoring scientists inside. The recorders had been instructed likewise. In the scoring room, two researchers obtained the clinical data. The Loe and Silness plaque - and gingival index were recorded on the mesial, buccal, distal and palatal aspects of teeth 16, 15, 14, 13 and 23, 24, 25, 26. Adverse events like discoloration observed during the clinical examination (yes/no) and clinically visible oral mucosal reactions were registered. In addition, plaque index by Quigley and Hine, the Turesky modification, was registered. All clinical registrations were performed by the same experienced periodontist, leaving her colleague to register recordings on specially designed charts. The clinical crew was kept blind to the group allocation of the participants at all times, as the only one that had access to the code-book was the statistician who did not participate in the clinical events.

Statistics The present experiment aimed at comparing the plaque and gingivitis preventing effect of the 0.12% - and 0.06% chlorhexidine solutions with the gold standard 0.2% chlorhexidine group.

The total number of participants was 60, with 20 participants in each group. The number of participants was based on the following power calculation. The power analysis was based on the variable 'average plaque score in each participant'. When comparing average plaque scores in two groups, a two-sided independent samples t-test was used, with 5% significance level. Average standard deviation in the 3 groups was 0.40. It may be shown that in order to have 80% test power to detect a mean difference in average plaque score of at least 0.40 between two groups, at least 15 participants must be included in each group. Because some drop-outs were expected, it was decided to include 60 subjects in the study. Because 80% test power is generally accepted as sufficiently high in clinical studies, and the mean difference in mesial plaque score between group 1 and group 3 was 0.41, the above calculation suggest that the study had acceptable test power.

When comparing mean plaque score in two groups, a two-sided independent sample t-test was used, with a 5% significance level. When comparing proportion of subjects with a particular adverse effect, the "linear by linear association chi-square" test was used. The statistical analysis was conducted using the software of Statistical Package for the Social Sciences (SPSS) for Windows, Version 16.0.

The distributions of the outcome variables were checked, and found to be sufficiently close to the normal distribution to allow for the use of a t-test.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking subjects,
* healthy subjects
* having at least three of the following teeth in maxillary right and left quadrant: the canine, 1st bicuspid, 2nd bicuspid, 1st molar,
* healthy gingiva and periodontium

Exclusion Criteria:

* pregnancy
* lactation
* any chronic diseases
* clinical signs or symptoms of acute infection in the oral cavity
* any prescribed or non-prescription systemic or topical medication except oral contraceptives
* use of systemic antibiotics the last 3 months prior to the start of the study history of alcohol or drug abuse
* participation in other clinical studies in the last 4 weeks.

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Estimated)
Dates: Start 2016-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Plaque index of Silness and Loe (PI) 1964 | 21 days
  0= No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  2. Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
  3. Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.

SECONDARY OUTCOMES:
Gingival index of Løe (GI) and Silness 1963 | 21 days
  0 No inflammation.
  1. Mild inflammation, slight change in color, slight edema, no bleeding on probing.
  2. Moderate inflammation, moderate glazing, redness, bleeding on probing.
  3. Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding.

OTHER OUTCOMES:
Side effects | 21 days
  All reported side subjective side effects like "taste perturbation" (Yes/No) "numbness" (Yes/No) "soar tongue tip" (Yes/No) "Mucosal ulcers" (yes/No)
subjective and objective discoloration of teeth | 21 days
  Discoloration of dental surfaces (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Hans R Preus, PhD, Principal Investigator — Department of periodontics, Dental Faculty, UiO
Locations (1):
- Department of Periodontology, Institute of Clinical Odontology, Dental Faculty, University of Oslo, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Yes
Via Scientific Journals

REFERENCES:
- [Background] Denton, G. W. Disinfection, Sterilization and Preservation, 4th ed, pp. 274-89.
- [Background] Loe H, Schiott CR. The effect of mouthrinses and topical application of chlorhexidine on the development of dental plaque and gingivitis in man. J Periodontal Res. 1970;5(2):79-83. doi: 10.1111/j.1600-0765.1970.tb00696.x. No abstract available. PMID 4254172
- [Background] Altman DG. Clinical trials. Practical statistics for medical research. London: Chapman & Hall/CRC; 1991. p 456.
- [Result] Davies A. The mode of action of chlorhexidine. J Periodontal Res Suppl. 1973;12:68-75. doi: 10.1111/j.1600-0765.1973.tb02167.x. No abstract available. PMID 4269603
- [Result] Gjermo P. Hibitane in periodontal disease. J Clin Periodontol. 1977 Dec;4(5):94-101. doi: 10.1111/j.1600-051x.1977.tb00055.x. No abstract available. PMID 275281
- [Result] Hull PS. Chemical inhibition of plaque. J Clin Periodontol. 1980 Dec;7(6):431-42. doi: 10.1111/j.1600-051x.1980.tb02150.x. PMID 7012186
- [Result] Addy M. Chlorhexidine compared with other locally delivered antimicrobials. A short review. J Clin Periodontol. 1986 Nov;13(10):957-64. doi: 10.1111/j.1600-051x.1986.tb01434.x. PMID 3540026
- [Result] Owens J, Addy M, Faulkner J, Lockwood C, Adair R. A short-term clinical study design to investigate the chemical plaque inhibitory properties of mouthrinses when used as adjuncts to toothpastes: applied to chlorhexidine. J Clin Periodontol. 1997 Oct;24(10):732-7. doi: 10.1111/j.1600-051x.1997.tb00190.x. PMID 9350557
- [Result] Gjermo P, Rolla G, Arskaug L. Effect on dental plaque formation and some in vitro properties of 12 bis-biguanides. J Periodontal Res Suppl. 1973;12:81-92. doi: 10.1111/j.1600-0765.1973.tb02169.x. No abstract available. PMID 4269606
- [Result] Berchier CE, Slot DE, Van der Weijden GA. The efficacy of 0.12% chlorhexidine mouthrinse compared with 0.2% on plaque accumulation and periodontal parameters: a systematic review. J Clin Periodontol. 2010 Sep;37(9):829-39. doi: 10.1111/j.1600-051X.2010.01575.x. Epub 2010 Jul 7. PMID 20618550
- [Result] QUIGLEY GA, HEIN JW. Comparative cleansing efficiency of manual and power brushing. J Am Dent Assoc. 1962 Jul;65:26-9. doi: 10.14219/jada.archive.1962.0184. No abstract available. PMID 14489483
- [Result] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376
- [Result] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Result] LOE H, THEILADE E, JENSEN SB. EXPERIMENTAL GINGIVITIS IN MAN. J Periodontol (1930). 1965 May-Jun;36:177-87. doi: 10.1902/jop.1965.36.3.177. No abstract available. PMID 14296927
- [Result] Preus HR, Aass AM, Hansen BF, Moe B, Gjermo P. A randomized, single-blind, parallel-group clinical study to evaluate the effect of soluble beta-1,3/1,6-glucan on experimental gingivitis in man. J Clin Periodontol. 2008 Mar;35(3):236-41. doi: 10.1111/j.1600-051X.2007.01183.x. PMID 18269662
- [Result] Preus HR, Koldsland OC, Aass AM, Sandvik L, Hansen BF. The plaque- and gingivitis-inhibiting capacity of a commercially available essential oil product. A parallel, split-mouth, single blind, randomized, placebo-controlled clinical study. Acta Odontol Scand. 2013 Nov;71(6):1613-9. doi: 10.3109/00016357.2013.782506. Epub 2013 May 3. PMID 23638764
- [Result] Harper PR, Milsom S, Wade W, Addy M, Moran J, Newcombe RG. An approach to efficacy screening of mouthrinses: studies on a group of French products (II). Inhibition of salivary bacteria and plaque in vivo. J Clin Periodontol. 1995 Sep;22(9):723-7. doi: 10.1111/j.1600-051x.1995.tb00833.x. PMID 7593704
- [Result] Keijser JA, Verkade H, Timmerman MF, Van der Weijden FA. Comparison of 2 commercially available chlorhexidine mouthrinses. J Periodontol. 2003 Feb;74(2):214-8. doi: 10.1902/jop.2003.74.2.214. PMID 12666710
- [Result] Franco Neto CA, Parolo CC, Rosing CK, Maltz M. Comparative analysis of the effect of two chlorhexidine mouthrinses on plaque accumulation and gingival bleeding. Braz Oral Res. 2008 Apr-Jun;22(2):139-44. doi: 10.1590/s1806-83242008000200008. PMID 18622483
- [Result] Pizzo G, Guiglia R, Imburgia M, Pizzo I, D'Angelo M, Giuliana G. The effects of antimicrobial sprays and mouthrinses on supragingival plaque regrowth: a comparative study. J Periodontol. 2006 Feb;77(2):248-56. doi: 10.1902/jop.2006.050116. PMID 16460251
- [Result] Quirynen M, Avontroodt P, Peeters W, Pauwels M, Coucke W, van Steenberghe D. Effect of different chlorhexidine formulations in mouthrinses on de novo plaque formation. J Clin Periodontol. 2001 Dec;28(12):1127-36. doi: 10.1034/j.1600-051x.2001.281207.x. PMID 11737510
- [Result] Smith RG, Moran J, Addy M, Doherty F, Newcombe RG. Comparative staining in vitro and plaque inhibitory properties in vivo of 0.12% and 0.2% chlorhexidine mouthrinses. J Clin Periodontol. 1995 Aug;22(8):613-7. doi: 10.1111/j.1600-051x.1995.tb00814.x. PMID 8583018
- [Result] Van Strydonck DA, Timmerman MF, van der Velden U, van der Weijden GA. Plaque inhibition of two commercially available chlorhexidine mouthrinses. J Clin Periodontol. 2005 Mar;32(3):305-9. doi: 10.1111/j.1600-051X.2005.00681.x. PMID 15766375
- [Result] 26. Valør LO, Norton IKR, Koldsland OC, Aass AM, Sandvik L, Preus HR. The plaque- and gingivitis inhibiting capacity of a commercially available mouthwash containing essential oils and ethyl lauroyl arginate. A parallel, split-mouth, double blind, randomized, placebo-controlled clinical study. In press
- [Result] Preus HR, Dahlen G, Gjermo P, Baelum V. Microbiologic Observations After Four Treatment Strategies Among Patients With Periodontitis Maintaining a High Standard of Oral Hygiene: Secondary Analysis of a Randomized Controlled Clinical Trial. J Periodontol. 2015 Jul;86(7):856-65. doi: 10.1902/jop.2015.140620. Epub 2015 Mar 12. PMID 25762359
- [Result] Vatne JF, Gjermo P, Sandvik L, Preus HR. Patients' perception of own efforts versus clinically observed outcomes of non-surgical periodontal therapy in a Norwegian population: an observational study. BMC Oral Health. 2015 May 17;15:61. doi: 10.1186/s12903-015-0037-3. PMID 25981528
- [Derived] Haydari M, Bardakci AG, Koldsland OC, Aass AM, Sandvik L, Preus HR. Comparing the effect of 0.06% -, 0.12% and 0.2% Chlorhexidine on plaque, bleeding and side effects in an experimental gingivitis model: a parallel group, double masked randomized clinical trial. BMC Oral Health. 2017 Aug 18;17(1):118. doi: 10.1186/s12903-017-0400-7. PMID 28821290